CLINICAL TRIAL: NCT07188116
Title: Correlation Between COVID-19 and Radiation Pneumonitis in Breast Cancer: A Historical Cohort Study
Brief Title: Correlation Between COVID-19 and Radiation Pneumonitis in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COBRA-001
Record Dates: First submitted 2025-09-22; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Radiation Pneumonia; COVID-19
Keywords: Retrospective Analysis; COVID-19; Radiation Pneumonitis; Propensity Score Matching; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Radiation Pneumonitis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without COVID-19: No COVID-19 infection
  Interventions: Other: COVID-19
- With COVID-19: With COVID-19 infection
  Interventions: Other: COVID-19

INTERVENTIONS:
Other: COVID-19 — The COVID-19 infection situation was used as an intervention measure, and the cohort was divided into groups.

SUMMARY:
This study was designed as a single-center retrospective analysis aimed at investigating whether COVID-19 infection increases the risk or burden of radiation-induced pneumonitis in breast cancer patients.

DETAILED DESCRIPTION:
This study was designed as a single-center retrospective analysis aimed at investigating whether COVID-19 infection increases the risk or burden of radiation-induced pneumonitis in breast cancer patients. Breast cancer patients who underwent radiotherapy at the Cancer Center of Zhejiang Hospital between January 1, 2021, and June 30, 2024, were screened for eligibility. Patients who met the inclusion criteria were identified through the hospital information system, and their clinical records were reviewed. Follow-up was conducted via telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

1. patients with pathologically or cytologically confirmed primary breast cancer,
2. aged 18 years or older but younger than 80 years,
3. with complete and reliable medical records,
4. for those with COVID-19 infection, documented evidence of a positive test result.

Exclusion Criteria:

1. concomitant pulmonary malignancies,
2. a history of prior thoracic radiotherapy,
3. concurrent pulmonary infections other than COVID-19 during radiotherapy,
4. missing key data with loss to follow-up,
5. or any other condition considered unsuitable for enrollment by the investigators.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who underwent radiotherapy at the Cancer Center of Zhejiang Hospital between January 1, 2021, and June 30, 2024, were screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiation Pneumonitis Situation | From January 2021 to June 2024
  The incidence rate, severity and onset time of radiation pneumonitis

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Hospital, Department of Oncology, Hangzhou, China, 310030, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No